CLINICAL TRIAL: NCT01754805
Title: A Phase 1b, Open-Label, Single Sequence, Drug Interaction Study to Evaluate the Pharmacokinetics of ASP015K and Methotrexate in Subjects With Rheumatoid Arthritis
Brief Title: A Drug Interaction Study to Evaluate the Pharmacokinetics of ASP015K and Methotrexate in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 015K-CL-PK13
Record Dates: First submitted 2012-12-19; First posted 2012-12-21 (Estimated); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Rheumatoid Arthritis
Keywords: ASP015K; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — peficitinib; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ASP015K and methotrexate (Experimental): Patients receive a single dose of methotrexate on day 1 and day 8 and ASP015K (twice daily) on days 3 through 8 plus the morning of day 9.
  Interventions: Drug: peficitinib; Drug: methotrexate

INTERVENTIONS:
Drug: peficitinib — oral
  Other Names: ASP015K
Drug: methotrexate — oral

SUMMARY:
A drug interaction study to evaluate the effect of ASP015K (twice daily) on the pharmacokinetics (PK) of once weekly oral methotrexate (MTX).

DETAILED DESCRIPTION:
Patients check in on day -1 and remain confined until all the exit procedures are performed on the morning of day 10. Patients to return for 1 post-treatment follow-up visit on day 13.

Patients receive a single dose of methotrexate on day 1 and day 8 and ASP015K (twice daily) on days 3 through 8 plus the morning of day 9.

ELIGIBILITY:
Inclusion Criteria:

1. If female, subject must be at least 2 years post menopausal or is surgically sterile per documentation provided by a medical professional and the subject is not pregnant as documented by a negative serum pregnancy test at Screening and negative urine pregnancy test at check-in
2. If male, subject must agree to sexual abstinence and/or to use a highly effective method of birth control during the study period and for 60 days after the last dose of study drug
3. Subject must have a clinical diagnosis of Rheumatoid Arthritis (RA) at least 6 months prior to Screening
4. Subject must be on a stable 15 - 25 mg dose of methotrexate > 28 days prior to Screening
5. If subject is on a non-biologic disease modifying anti-rheumatic drug (DMARDs) therapy, the dose must be stable > 28 days prior to Screening
6. Subject must be willing and able to comply with the study requirements

Exclusion Criteria:

1. Subject has a previous history of any clinically significant neurological, gastrointestinal, renal, hepatic, pulmonary, metabolic, cardiovascular, psychiatric, endocrine, hematological disorder or disease, or any other medical condition that would preclude participation in the study
2. Subject has a known history of positive test for hepatitis B surface antigen (HbsAg) or hepatitis C antibody or history of a positive test for human immunodeficiency virus (HIV) infection
3. Subject has received live virus vaccination within the last 30 days prior to study drug administration
4. Subject has a Body Mass Index (BMI) > 35 (kg/m2)
5. Subject is on biologic disease modifying anti-rheumatic drug (DMARDs) therapy
6. Subject has a current history of anemia as defined by hemoglobin of less than 12 g/dL
7. Subject has a recent history (within the last 6 months) of drug or alcohol abuse or a positive urine screen for alcohol or drugs of abuse/illegal drugs at Screening or check-in
8. Subject has received any investigational agent within 30 days of screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-01-22 (Actual); Primary Completion 2010-03-25 (Actual); Study Completion 2010-03-25 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of methotrexate (MTX): Area under the concentration-time curve from time of dosing to infinity (AUCinf) | Days 1 and 8
Pharmacokinetics of methotrexate (MTX): Maximum concentration (Cmax) | Days 1 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Global Development
Locations (1):
- Anniston, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Zhu T, Moy S, Valluri U, Cao Y, Zhang W, Sawamoto T, Chindalore V, Akinlade B. Investigation of Potential Drug-Drug Interactions between Peficitinib (ASP015K) and Methotrexate in Patients with Rheumatoid Arthritis. Clin Drug Investig. 2020 Sep;40(9):827-838. doi: 10.1007/s40261-020-00937-z. PMID 32591978
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=325